CLINICAL TRIAL: NCT01266018
Title: Phase II Study of ADI-PEG 20 in Patients With Relapsed Sensitive or Refractory Small Cell Lung Cancer
Brief Title: Study of ADI-PEG 20 in Patients With Relapsed Sensitive or Refractory Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy in Cohort 2; slow enrollment in Cohort 1
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Duke University (Other); St. Bartholomew's Hospital (Other); Krankenhaus Nordwest (Other); Saint-Luc University Hospital (Unknown); National Taiwan University Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other); Austin Health (Other Government); Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2009-007; Pro00022622 (Other: Duke University Medical Center)
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; SCLC; ADI-PEG 20; arginine deiminase pegylated
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Sensitive Disease (Experimental): Cohort 1 comprised subjects with "sensitive" disease, defined as subjects who were treated with 1 previous line of chemotherapy and maintained an appropriate response for 90 days or more. Subjects received 4 administrations of ADI-PEG 20 (320 IU/m^2) followed by 1 week of follow-up in each treatment cycle.
  Interventions: Drug: ADI-PEG 20 (Arginine deiminase pegylated)
- Cohort 2: Refractory Disease (Experimental): Cohort 2 comprised subjects with "refractory" disease, defined as subjects who either (a) were treated with 1 previous line of chemotherapy and either had no response or progressed < 90 days after completing treatment or (b) required third-line therapy, i.e., had completed 2 previous lines of chemotherapy, regardless of response. Subjects received 4 administrations of ADI-PEG 20 (320 IU/m^2) followed by 1 week of follow-up in each treatment cycle.
  Interventions: Drug: ADI-PEG 20 (Arginine deiminase pegylated)

INTERVENTIONS:
Drug: ADI-PEG 20 (Arginine deiminase pegylated) — ADI-PEG 20 was administered intramuscularly (IM) at a fixed dose of 320 IU/m^2 (36.8 mg/m^2) once weekly for 4 weeks followed by a 1-week follow-up (1 cycle)
  Other Names: ADI; Arginine deiminase pegylated

SUMMARY:
This was a 2-arm, open-label, phase 2 study of pegylated arginine deiminase (ADI-PEG) 20 in subjects with relapsed sensitive or refractory small cell lung cancer (SCLC). ADI-PEG 20 was administered intramuscularly (IM) at a fixed dose of 320 IU/m^2 once weekly for a 4-week cycle. The primary objective was to assess clinical efficacy with a primary endpoint of tumor response by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after 4 weeks. Secondary objectives were to assess the safety, pharmacodynamics, and immunogenicity of ADI-PEG 20, as well as clinical efficacy with a secondary endpoint of overall survival.

DETAILED DESCRIPTION:
Subjects were enrolled sequentially (non-randomized) into two separate cohorts in parallel. Cohort 1 comprised subjects with "sensitive" disease and Cohort 2 comprised subjects with "refractory" disease. Both cohorts received the same treatment regimen consisting of 4 weekly IM administrations of ADI-PEG 20 (320 IU/m^2), followed by a 1-week follow-up (1 cycle). No dose adjustment was allowed. Additional treatment cycles were permitted in the absence of disease progression requiring other therapeutic interventions.

Each cohort was to be enrolled in 2 stages. In the first stage, 15 subjects were to be accrued in Cohort 1 and 12 subjects in Cohort 2. If ≥ 3 subjects met the primary endpoint in Cohort 1, then an additional 13 subjects were to be accrued in the second stage. If ≤ 2 subjects met the primary endpoint in Cohort 1, then the study was to be terminated and declared negative for Cohort 1. If ≥ 1 subject met the primary endpoint in Cohort 2, then an additional 4 subjects were to be accrued in the second stage. If no subjects met the primary endpoint in Cohort 2, then the study was to be terminated and declared negative. Additionally, if at any time a death or two grade 4 adverse events (AEs) that were definitely related or probably related to the study drug occurred, then the study was to be stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have had histologically documented SCLC
2. Assigned to one of two cohorts based on the following characteristics: Cohort 1: "Sensitive" disease subjects who had 1 previous line of chemotherapy and maintained an appropriate response for 90 days or more; or Cohort 2: "Refractory" disease subjects, who had (a) 1 previous line of chemotherapy and either had no response or progressed in less than 90 days after completing treatment or (b) any subject ("sensitive" or "refractory") in need of third-line therapy, i.e., who completed or failed 2 previous lines of chemotherapy
3. Measurable disease using RECIST version 1.1
4. Argininosuccinate synthetase (ASS) tumor expression was either negative or < 5% + tumor cells by immunohistochemistry analysis
5. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2
6. Laboratory parameters for vital functions in the normal range. Laboratory abnormalities that were not clinically significant were generally permitted, except for the following laboratory parameters, which were to be within the ranges specified:

   * Neutrophil count: ≥ 1.5 x 10^9/L
   * Lymphocyte count: ≥ 0.5 x 10^9/L
   * Platelet count: ≥ 50 x 10^9/L
   * Serum creatinine: ≤ 1.5 x upper limit of normal (ULN) (or creatinine clearance ≥ 60 mL/min)
   * Serum bilirubin: ≤ 2 mg/dL (or ≤ 34 µmol/L)
   * Serum uric acid: ≤ 8 mg/dL (or ≤ 0.48 mmol/L)
   * International normalized ratio (INR): ≤ 1.5
   * Partial thromboplastin time: ≤ 1.5 x ULN
7. Age ≥ 18 years
8. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Previous treatment with ADI-PEG 20
2. Known allergy to pegylated products
3. History of uncontrolled seizures
4. Serious illnesses, e.g., serious infections requiring antibiotics, bleeding disorders, or any condition that in the opinion of the Investigator would interfere with the ability of the patient to fulfill the study requirements
5. Metastatic disease to the central nervous system, unless treated and stable
6. Known immunodeficiency or human immunodeficiency virus (HIV) positivity
7. Participation in another clinical trial involving another investigational agent within 3 weeks prior to first dosing of study agent
8. Any other malignancy that required protocol-specified restricted concomitant therapy
9. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study
10. Lack of availability for clinical follow-up assessment
11. Pregnancy or breast feeding
12. Refusal or inability to use effective means of contraception for men and women of childbearing potential for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Krug, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
- University Clinic Saint-Luc, Brussels, Belgium
- Krankenhaus Nordwest, Frankfurt, Germany
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - LinKou Branch, Taoyuan District
- St. Bartholomew's Hospital, West Smithfield, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Sensitive Disease: Cohort 1 comprised subjects with "sensitive" disease, defined as subjects who were treated with 1 previous line of chemotherapy and maintained an appropriate response for 90 days or more.
- Cohort 2: Refractory Disease: Cohort 2 comprised subjects with "refractory" disease, defined as subjects who either (a) were treated with 1 previous line of chemotherapy and either had no response or progressed < 90 days after completing treatment or (b) required third-line therapy, i.e., had completed 2 previous lines of chemotherapy, regardless of response
Period: Overall Study
Arm/Group | Cohort 1: Sensitive Disease | Cohort 2: Refractory Disease
Started | 9 | 13
Completed | 8 (Defined as evaluable for the primary endpoint) | 12
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Progressive disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- All Enrolled Subjects: Includes all subjects enrolled in Cohort 1 (n = 9) and Cohort 2 (n = 13).
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 1
  United States | 11
  Taiwan | 6
  United Kingdom | 3
  Germany | 1
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (5.6)
Argininosuccinate Synthetase (ASS) Assay Result [Number; unit: participants] — ASS tumor expression was either negative or < 5% positive tumor cells by immunohistochemistry
  participants
    Negative | 11
    <5% cells positive | 11

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Tumor responses were evaluated using any appropriate imaging type and were categorized according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Per RECIST for target lesions and assessed by MRI:
  Complete Response (CR): Disappearance of all target lesions [no evidence of disease]; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Every 4 to 8 weeks for up to 16 weeks
Population: Includes all patients who were evaluable for tumor response allocation.
Measure: Number; unit: participants
Groups:
- Cohort 1: Sensitive Disease: Includes subjects with "sensitive" disease, defined as subjects who were treated with 1 previous line of chemotherapy and maintained an appropriate response for 90 days or more.
- Cohort 2: Refractory Disease: Includes subjects with "refractory" disease, defined as subjects who either (a) were treated with 1 previous line of chemotherapy and either had no response or progressed < 90 days after completing treatment or (b) required third-line therapy, i.e., had completed 2 previous lines of chemotherapy, regardless of response.
Arm/Group | Cohort 1: Sensitive Disease | Cohort 2: Refractory Disease
Number analyzed (Participants) | 8 | 12
participants
  Stable disease | 2 | 2
  Progressive disease | 6 | 10

2. Secondary Outcome: Assessment of Safety of Arginine Deiminase Pegylated (ADI-PEG) 20
Description: Analysis of treatment-emergent adverse events (TEAEs) reported from clinical laboratory tests, physical examinations, and vital signs.
Time Frame: Every 1 to 4 weeks for up to 16 weeks
Population: The Safety Analysis Set comprises all subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Sensitive Disease | Cohort 2: Refractory Disease
Number analyzed (Participants) | 9 | 13
participants
  Any TEAE | 9 | 12
  Grade 3 TEAE | 5 | 1
  Grade 4 TEAE | 1 | 2
  Grade 5 TEAE (Death) | 0 | 3
  Treatment-related TEAE | 4 | 7
  Serious TEAE | 5 | 5
  TEAE leading to withdrawal | 0 | 3

3. Secondary Outcome: Assessment of Pharmacodynamics of ADI-PEG 20
Description: Blood samples were collected from all subjects at enrollment, prior to each treatment, and at the end of study to evaluate changes in plasma arginine and citrulline levels following administration of ADI-PEG 20. Disease state (ie, relapsed sensitive vs refractory) was not considered relevant to this analysis and as such samples were collected without regard for cohort assignment.
Time Frame: Every 1 to 4 weeks for up to 16 weeks
Population: The Pharmacodynamic Analysis Set comprises all subjects who received at least 1 dose of study drug and provided plasma samples for pharmacodynamic analyses. A total of 121 plasma samples from 21 subjects were analyzed. Summary data are presented through Day 58, i.e., the last time point with at least 3 samples available for calculation of a mean.
Measure: Mean (Full Range); unit: uM
Groups:
- All Subjects (Pharmacodynamic Analysis Set): Includes all subjects in Cohort 1 (n = 9) and Cohort 2 (n = 12) who received at least 1 dose of study drug and provided plasma samples for pharmacodynamic analyses.
Arm/Group | All Subjects (Pharmacodynamic Analysis Set)
Number analyzed (Participants) | 21
uM
  Arginine (Day 0) | 69 [39 to 96]
  Arginine (Day 1) | 110 [26 to 321]
  Arginine (Day 8) | 2 [1 to 5]
  Arginine (Day 15) | 2 [1 to 5]
  Arginine (Day 22) | 3 [1 to 12]
  Arginine (Day 29) | 2 [1 to 5]
  Arginine (Day 36) | 16 [1 to 105]
  Arginine (Day 43) | 11 [1 to 67]
  Arginine (Day 50) | 29 [1 to 69]
  Arginine (Day 58) | 52 [1 to 113]
  Citrulline (Day 0) | 26 [14 to 40]
  Citrulline (Day 1) | 46 [9 to 232]
  Citrulline (Day 8) | 546 [91 to 912]
  Citrulline (Day 15) | 684 [136 to 1190]
  Citrulline (Day 22) | 495 [71 to 1130]
  Citrulline (Day 29) | 409 [91 to 982]
  Citrulline (Day 36) | 223 [15 to 367]
  Citrulline (Day 43) | 222 [60 to 530]
  Citrulline (Day 50) | 222 [42 to 632]
  Citrulline (Day 58) | 119 [43 to 316]

4. Secondary Outcome: Assessment of Immunogenicity of ADI-PEG 20
Description: Blood samples were collected for all subjects at enrollment, prior to each treatment, and at the end of study to evaluate changes in ADI-PEG 20 antibody titer in peripheral blood over time. Disease state (ie, relapsed sensitive vs refractory) was not considered relevant to this analysis and as such samples were collected without regard for cohort assignment.
Time Frame: Every 1 to 4 weeks for up to 16 weeks
Population: as for outcome 3
Measure: Mean (Full Range); unit: log 10 IU/mL
Arm/Group | All Subjects (Pharmacodynamic Analysis Set)
Number analyzed (Participants) | 21
log 10 IU/mL
  Antibody titer (Day 0) | 0.7 [0 to 2]
  Antibody titer (Day 1) | 0.5 [0 to 2]
  Antibody titer (Day 8) | 0.4 [0 to 2]
  Antibody titer (Day 15) | 1.4 [0 to 3]
  Antibody titer (Day 22) | 1.5 [0 to 4]
  Antibody titer (Day 29) | 1.3 [0 to 3]
  Antibody titer (Day 36) | 1.9 [0 to 5]
  Antibody titer (Day 43) | 2.2 [0 to 4]
  Antibody titer (Day 50) | 3.4 [1 to 6]
  Antibody titer (Day 58) | 4.0 [3 to 5]

5. Secondary Outcome: Assessment of Overall Survival
Description: Overall survival was measured from the initial date of treatment to the recorded date of death. Because the study was terminated prematurely, no statistical analyses of overall survival data were performed.
Time Frame: Every 4 weeks for up to 16 months
Population: Subjects who had survival status recorded during post-study follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Sensitive Disease | Cohort 2: Refractory Disease
Number analyzed (Participants) | 6 | 11
Participants
  Alive at last follow-up | 4 | 4
  Not alive at last follow-up | 2 | 7

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs).
Description: AE documentation included onset/resolution dates, severity using NCI CTCAE (v4.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per subject at the maximum reported grade.
Groups:
- All Subjects (Safety Analysis Set): Includes all subjects in Cohort 1 (n = 9) and Cohort 2 (n = 13) who received at least 1 dose of study drug.
Arm/Group | All Subjects (Safety Analysis Set)
Serious Adverse Events (participants affected / at risk) | 10/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (Safety Analysis Set) (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (Safety Analysis Set) (N=22)
Tachycardia (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 10
Asthenia (General disorders) | 4
Chest discomfort (General disorders) | 2
Lower respiratory tract infection (Infections and infestations) | 2
White blood cell count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 3
Blood creatinine increased (Investigations) | 2
Haemoglobin decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of efficacy and slow enrollment; therefore, only 22 of the planned 45 subjects were enrolled, treated, and evaluated for study endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less